CLINICAL TRIAL: NCT04334291
Title: International COVID19 Clinical Evaluation Registry: HOPECOVID19. (Health Outcome Predictive Evaluation for COVID19)
Brief Title: International COVID19 Clinical Evaluation Registry,
Acronym: HOPE COVID 19
Status: Completed | Type: Observational
Sponsor: IVAN J NUÑEZ GIL (Other)
Responsible Party: Sponsor-Investigator, IVAN J NUÑEZ GIL, Principal Investigator. Attending Physician. MD, PhD, FESC, St Carlos Hospital, Madrid, Spain
Organization: St Carlos Hospital, Madrid, Spain (Other)
Other Study IDs: 20/241-E; EUPAS34399 (Other: EMA)
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Observational (registry) — Observational study.

SUMMARY:
The investigators propose to select all COVID 19 patients attended in any health center (with in hospital beds), who have been discharged or have died at the time of the evaluation.

The main objective of the present study is to carefully characterize the clinical profile of patients infected with COVID-19 in order to develop a simple prognostic clinical score allowing, in selected cases, rapid logistic decision making (discharge with follow-up, referral to provisional/field hospitals or admission to more complex hospital centers).

As secondary objectives, the analysis of the risk-adjusted influence of treatments and previous comorbidities of patients infected with the disease will be performed.

DETAILED DESCRIPTION:
INTRODUCTION. The disease caused by the new respiratory virus (coronavirus) designated as SARS-CoV-2 has recently been classified as a pandemic by the WHO.

With an increasing number of confirmed cases in most countries worldwide, it is responsible for a significant morbidity and mortality and has motivated the implementation of measures at national and international levels with a great impact on the way of life of people throughout the whole planet.

In addition, this condition currently threatens many countries with the collapse of health systems, producing serious logistical problems due to extensive affectation of the population, which can worsen the prognosis of those primarily affected by COVID 19 and other patients with different pathologies and who may have difficulties to get healthcare.

Limited clinical information is available and generally limited to the Asian population, since the first cases were identified in Wuhan (Hubei, China).

PURPOSE. The main objective of the present study is to carefully characterize the clinical profile of patients infected with COVID-19 in order to develop a simple prognostic clinical score allowing, in selected cases, rapid logistic decision making (discharge with follow-up, referral to provisional/field hospitals or admission to more complex hospital centers).

As secondary objectives, the analysis of the risk-adjusted influence of treatments (ie. ACEIs, ARBs) and previous comorbidities of patients infected with the disease will be performed.

DESIGN AND STATISTICAL ANALYSIS Cross-sectional and ambispective registry, a real life "all comers" type, with voluntary participation, without funding or conflicts of interest. It is a study initiated by researcher that will have advanced statistical support from the IMAS foundation (Institute for the Improvement of Health Care, Madrid, Spain), that will serve as statistical core.

International level.

PARTICIPANTS PROTOCOL. The study has been approved by Hospital Clinico San Carlos Ethic´s Committee (20/241-E) and the institutional board of each participating center. It has received an AEMPS classification (EPA-0D).

The researchers aimto select all the patients attended in any health center (with in hospital beds), who have been discharged or have died at the time of the evaluation.

All will be considered eligible with a positive COVID 19 test (any type) or if their attending physicians consider them highly likely to have presented the infection.

Given the anonymous characteristics of the registry and the health alarm situation generated by the virus, in principle, it is not considered necessary to provide written informed consent.

- Inclusion criteria Patients discharged (deceased or alive) from any hospital center with a confirmed diagnosis or a COVID-19 high suspicion.

There are no exclusion criteria, except for the patient's explicit refusal to participate.

DATA BASE. An anonymized database is presented in electronic format, to be filled in at each participating center (www.HopeProjectMD.com).

In theory, all information could be obtained from electronic records (medical history).

If deemed necessary, the investigator may call patients in order to establish their vital status (strongly warranted), as well as the results of the RNA test (or antibody) , if they were pending during their stay.

SAMPLE SIZE. It would not be possible to estimate for the sample size based on literature reports. Thus, HOPE will aim to get the maximum numbers of patients possible.

OUTCOMES. Primary: All-cause mortality. The major contributors of increased mortality will be assessed.

Secondary: In stay events, defined by the attending physician.

* In hospital stay.
* Heart failure.
* Renal failure.
* Respiratory Insufficiency.
* Upper respiratory tract involvement.
* Pneumonia.
* Sepsis.
* Systemic inflammatory response Syndrome.
* Clinically relevant bleeding.
* Hemoptysis.
* Embolic event
* Other complications.
* Causes of death. Depending the results of the main interim analysis, the main DB could be slightly modified and several sub analyses could be proposed after sensitivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged (deceased or alive) from any hospital center with a confirmed diagnosis or a COVID-19 high suspicion.

Exclusion Criteria:

* There are no exclusion criteria, except for the patient's explicit refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed diagnosis or a COVID-19 high suspicion.
Sampling Method: Non-Probability Sample
Enrollment: 8168 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Death | through study completion, an average of 1 month
  All cause

SECONDARY OUTCOMES:
In hospital stay. | through study completion, an average of 1 month
  Days
Heart failure | through study completion, an average of 1 month
  According the attending physician.
Renal failure | through study completion, an average of 1 month
  According the attending physician.
Respiratory Insufficiency. | through study completion, an average of 1 month
  According the attending physician.
Upper respiratory tract involvement | through study completion, an average of 1 month
  According the attending physician.
Pneumonia | through study completion, an average of 1 month
  According the attending physician.
Sepsis | through study completion, an average of 1 month
  According the attending physician.
Systemic inflammatory response Syndrome. | through study completion, an average of 1 month
  According the attending physician.
Clinically relevant bleeding | through study completion, an average of 1 month
  According the attending physician.
Other complications. | through study completion, an average of 1 month
  According the attending physician.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Lclinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
IPD are to be share among HOPE researchers. However, the HOPE Steering committee is open to collaborative proposals.

REFERENCES:
- [Background] Nunez-Gil IJ, Estrada V, Fernandez-Perez C, Feltes G, Vedia O, Vergara-Uzcategui CE, Moreno-Menguia VH, Cerrato E, D'Ascenzo F, Raposeiras-Roubin S, Martin-Sanchez FJ, Alfonso-Rodriguez E, Huang J, Ramakrishna H, Gil-Higes E, Fernandez-Ortiz A, Macaya C. Health Outcome Predictive Evaluation for COVID 19 international registry (HOPE COVID-19), rationale and design. Contemp Clin Trials Commun. 2020 Dec;20:100654. doi: 10.1016/j.conctc.2020.100654. Epub 2020 Sep 23. PMID 32989425
- [Background] Uribarri A, Nunez-Gil IJ, Aparisi A, Arroyo-Espliguero R, Maroun Eid C, Romero R, Becerra-Munoz VM, Feltes G, Molina M, Garcia-Aguado M, Cerrato E, Capel-Astrua T, Alfonso-Rodriguez E, Castro-Mejia AF, Raposeiras-Roubin S, Espejo C, Perez-Sole N, Bardaji A, Marin F, Fabregat-Andres O, D'ascenzo F, Santoro F, Akin I, Estrada V, Fernandez-Ortiz A, Macaya C; HOPE COVID-19 investigators. Atrial fibrillation in patients with COVID-19. Usefulness of the CHA2DS2-VASc score: an analysis of the international HOPE COVID-19 registry. Rev Esp Cardiol (Engl Ed). 2021 Jul;74(7):608-615. doi: 10.1016/j.rec.2020.12.009. Epub 2021 Jan 13. PMID 33583755
- [Background] Pepe M, Maroun-Eid C, Romero R, Arroyo-Espliguero R, Fernandez-Rozas I, Aparisi A, Becerra-Munoz VM, Garcia Aguado M, Brindicci G, Huang J, Alfonso-Rodriguez E, Castro-Mejia AF, Favretto S, Cerrato E, Albiol P, Raposeiras-Roubin S, Vedia O, Feltes Guzman G, Carrero-Fernandez A, Perez Cimarra C, Buzon L, Jativa Mendez JL, Abumayyaleh M, Corbi-Pascual M, Macaya C, Estrada V, Nestola PL, Biondi-Zoccai G, Nunez-Gil IJ. Clinical presentation, therapeutic approach, and outcome of young patients admitted for COVID-19, with respect to the elderly counterpart. Clin Exp Med. 2021 May;21(2):249-268. doi: 10.1007/s10238-021-00684-1. Epub 2021 Feb 8. PMID 33555436
- [Result] Rivera-Caravaca JM, Nunez-Gil IJ, Vivas D, Viana-Llamas MC, Uribarri A, Becerra-Munoz VM, Trabattoni D, Fernandez Rozas I, Feltes G, Lopez-Pais J, El-Battrawy I, Macaya C, Fernandez-Ortiz A, Estrada V, Marin F; HOPE COVID-19 Investigators. Clinical profile and prognosis in patients on oral anticoagulation before admission for COVID-19. Eur J Clin Invest. 2021 Jan;51(1):e13436. doi: 10.1111/eci.13436. Epub 2020 Nov 7. PMID 33080051
- [Result] Nunez-Gil IJ, Fernandez-Perez C, Estrada V, Becerra-Munoz VM, El-Battrawy I, Uribarri A, Fernandez-Rozas I, Feltes G, Viana-Llamas MC, Trabattoni D, Lopez-Pais J, Pepe M, Romero R, Castro-Mejia AF, Cerrato E, Astrua TC, D'Ascenzo F, Fabregat-Andres O, Moreu J, Guerra F, Signes-Costa J, Marin F, Buosenso D, Bardaji A, Raposeiras-Roubin S, Elola J, Molino A, Gomez-Doblas JJ, Abumayyaleh M, Aparisi A, Molina M, Guerri A, Arroyo-Espliguero R, Assanelli E, Mapelli M, Garcia-Acuna JM, Brindicci G, Manzone E, Ortega-Armas ME, Bianco M, Trung CP, Nunez MJ, Castellanos-Lluch C, Garcia-Vazquez E, Cabello-Clotet N, Jamhour-Chelh K, Tellez MJ, Fernandez-Ortiz A, Macaya C; HOPE COVID-19 Investigators. Mortality risk assessment in Spain and Italy, insights of the HOPE COVID-19 registry. Intern Emerg Med. 2021 Jun;16(4):957-966. doi: 10.1007/s11739-020-02543-5. Epub 2020 Nov 9. PMID 33165755
- [Result] Nunez-Gil IJ, Estrada V, Fernandez-Perez C, Fernandez-Rozas I, Martin-Sanchez FJ, Macaya C. The COVID-19 curve, health system overload, and mortality. Emergencias. 2020 Ago;32(4):293-295. No abstract available. English, Spanish. PMID 32692012
- [Result] Uribarri A, Nunez-Gil IJ, Aparisi A, Becerra-Munoz VM, Feltes G, Trabattoni D, Fernandez-Rozas I, Viana-Llamas MC, Pepe M, Cerrato E, Capel-Astrua T, Romero R, Castro-Mejia AF, El-Battrawy I, Lopez-Pais J, D'Ascenzo F, Fabregat-Andres O, Bardaji A, Raposeiras-Roubin S, Marin F, Fernandez-Ortiz A, Macaya C, Estrada V; HOPE COVID-19 Investigators. Impact of renal function on admission in COVID-19 patients: an analysis of the international HOPE COVID-19 (Health Outcome Predictive Evaluation for COVID 19) Registry. J Nephrol. 2020 Aug;33(4):737-745. doi: 10.1007/s40620-020-00790-5. Epub 2020 Jun 29. PMID 32602006
- [Result] Nunez-Gil IJ, Fernandez-Ortiz A, Maroud Eid C, Huang J, Romero R, Becerra-Munoz VM, Uribarri A, Feltes G, Trabatoni D, Fernandez-Rozas I, Viana-Llamas MC, Pepe M, Cerrato E, Bertaina M, Capel Astrua T, Alfonso E, Castro-Mejia AF, Raposeiras-Roubin S, D'Ascenzo F, Espejo Paeres C, Signes-Costa J, Bardaji A, Fernandez-Perez C, Marin F, Fabregat-Andres O, Akin I, Estrada V, Macaya C. Underlying heart diseases and acute COVID-19 outcomes. Cardiol J. 2021;28(2):202-214. doi: 10.5603/CJ.a2020.0183. Epub 2020 Dec 21. PMID 33346365
- [Result] Becerra-Munoz VM, Nunez-Gil IJ, Eid CM, Garcia Aguado M, Romero R, Huang J, Mulet A, Ugo F, Rametta F, Liebetrau C, Aparisi A, Fernandez-Rozas I, Viana-Llamas MC, Feltes G, Pepe M, Moreno-Rondon LA, Cerrato E, Raposeiras-Roubin S, Alfonso E, Carrero-Fernandez A, Buzon-Martin L, Abumayyaleh M, Gonzalez A, Fernandez Ortiz A, Macaya C, Estrada V, Fernandez-Perez C, Gomez-Doblas JJ. Clinical profile and predictors of in-hospital mortality among older patients hospitalised for COVID-19. Age Ageing. 2021 Feb 26;50(2):326-334. doi: 10.1093/ageing/afaa258. PMID 33201181
- [Result] Ruiz-Sanchez JG, Nunez-Gil IJ, Cuesta M, Rubio MA, Maroun-Eid C, Arroyo-Espliguero R, Romero R, Becerra-Munoz VM, Uribarri A, Feltes G, Trabattoni D, Molina M, Garcia Aguado M, Pepe M, Cerrato E, Alfonso E, Castro Mejia AF, Roubin SR, Buzon L, Bondia E, Marin F, Lopez Pais J, Abumayyaleh M, D'Ascenzo F, Rondano E, Huang J, Fernandez-Perez C, Macaya C, de Miguel Novoa P, Calle-Pascual AL, Estrada Perez V, Runkle I; HOPE COVID-19 investigators. Prognostic Impact of Hyponatremia and Hypernatremia in COVID-19 Pneumonia. A HOPE-COVID-19 (Health Outcome Predictive Evaluation for COVID-19) Registry Analysis. Front Endocrinol (Lausanne). 2020 Nov 30;11:599255. doi: 10.3389/fendo.2020.599255. eCollection 2020. PMID 33329400
- [Result] El-Battrawy I, Nunez-Gil IJ, Abumayyaleh M, Estrada V, Manuel Becerra-Munoz V, Uribarri A, Fernandez-Rozas I, Feltes G, Arroyo-Espliguero R, Trabattoni D, Lopez-Pais J, Pepe M, Romero R, Castro-Mejia AF, Cerrato E, Capel Astrua T, D'Ascenzo F, Fabregat-Andres O, Signes-Costa J, Marin F, Buonsenso D, Bardaji A, Jesus Tellez M, Fernandez-Ortiz A, Macaya C, Akin I. COVID-19 and the impact of arterial hypertension-An analysis of the international HOPE COVID-19 Registry (Italy-Spain-Germany). Eur J Clin Invest. 2021 Nov;51(11):e13582. doi: 10.1111/eci.13582. Epub 2021 Aug 19. PMID 34409593
- [Result] Signes-Costa J, Nunez-Gil IJ, Soriano JB, Arroyo-Espliguero R, Eid CM, Romero R, Uribarri A, Fernandez-Rozas I, Aguado MG, Becerra-Munoz VM, Huang J, Pepe M, Cerrato E, Raposeiras S, Gonzalez A, Franco-Leon F, Wang L, Alfonso E, Ugo F, Garcia-Prieto JF, Feltes G, Abumayyaleh M, Espejo-Paeres C, Jativa J, Masjuan AL, Macaya C, Carbonell Asins JA, Estrada V; HOPE COVID-19 investigators. Prevalence and 30-Day Mortality in Hospitalized Patients With Covid-19 and Prior Lung Diseases. Arch Bronconeumol. 2021 Apr;57:13-20. doi: 10.1016/j.arbres.2020.11.012. Epub 2020 Dec 16. PMID 34629634
- [Result] Santoro F, Nunez-Gil IJ, Vitale E, Viana-Llamas MC, Reche-Martinez B, Romero-Pareja R, Feltez Guzman G, Fernandez Rozas I, Uribarri A, Becerra-Munoz VM, Alfonso-Rodriguez E, Garcia-Aguado M, Huang J, Ortega-Armas ME, Garcia Prieto JF, Corral Rubio EM, Ugo F, Bianco M, Mulet A, Raposeiras-Roubin S, Jativa Mendez JL, Espejo Paeres C, Albarran AR, Marin F, Guerra F, Akin I, Cortese B, Ramakrishna H, Macaya C, Fernandez-Ortiz A, Brunetti ND. Antiplatelet therapy and outcome in COVID-19: the Health Outcome Predictive Evaluation Registry. Heart. 2022 Jan;108(2):130-136. doi: 10.1136/heartjnl-2021-319552. Epub 2021 Oct 5. PMID 34611045
- [Result] Nunez-Gil IJ, Olier I, Feltes G, Viana-Llamas MC, Maroun-Eid C, Romero R, Fernandez-Rozas I, Uribarri A, Becerra-Munoz VM, Alfonso-Rodriguez E, Garcia-Aguado M, Elola J, Castro-Mejia A, Pepe M, Garcia-Prieto JF, Gonzalez A, Ugo F, Cerrato E, Bondia E, Raposeiras-Roubin S, Mendez JLJ, Espejo C, Lopez-Masjuan A, Marin F, Lopez-Pais J, Abumayyaleh M, Corbi-Pascual M, Liebetrau C, Ramakrishna H, Estrada V, Macaya C, Fernandez-Ortiz A; HOPE COVID-19 Investigators (Cols Appendix). Renin-angiotensin system inhibitors effect before and during hospitalization in COVID-19 outcomes: Final analysis of the international HOPE COVID-19 (Health Outcome Predictive Evaluation for COVID-19) registry. Am Heart J. 2021 Jul;237:104-115. doi: 10.1016/j.ahj.2021.04.001. Epub 2021 Apr 15. PMID 33845032
- [Result] Porta-Etessam J, Nunez-Gil IJ, Gonzalez Garcia N, Fernandez-Perez C, Viana-Llamas MC, Eid CM, Romero R, Molina M, Uribarri A, Becerra-Munoz VM, Aguado MG, Huang J, Rondano E, Cerrato E, Alfonso E, Mejia AFC, Marin F, Roubin SR, Pepe M, Feltes G, Mate P, Cortese B, Buzon L, Mendez JJ, Estrada V. COVID-19 anosmia and gustatory symptoms as a prognosis factor: a subanalysis of the HOPE COVID-19 (Health Outcome Predictive Evaluation for COVID-19) registry. Infection. 2021 Aug;49(4):677-684. doi: 10.1007/s15010-021-01587-9. Epub 2021 Mar 1. PMID 33646505
- [Result] Espejo-Paeres C, Nunez-Gil IJ, Estrada V, Fernandez-Perez C, Uribe-Heredia G, Cabre-Verdiell C, Uribarri A, Romero R, Garcia-Aguado M, Fernandez-Rozas I, Becerra-Munoz V, Pepe M, Cerrato E, Raposeiras-Roubin S, Barrionuevo-Ramos M, Aveiga-Ligua F, Aguilar-Andrea C, Alfonso-Rodriguez E, Ugo F, Garcia-Prieto JF, Feltes G, Akin I, Huang J, Jativa J, Fernandez-Ortiz A, Macaya C, Carrero-Fernandez A, Signes-Costa J. Impact of smoking on COVID-19 outcomes: a HOPE Registry subanalysis. BMJ Nutr Prev Health. 2021 Jun 17;4(1):285-292. doi: 10.1136/bmjnph-2021-000269. eCollection 2021. PMID 34308137
- [Result] Viana-Llamas MC, Arroyo-Espliguero R, Silva-Obregon JA, Uribe-Heredia G, Nunez-Gil I, Garcia-Magallon B, Toran-Martinez CG, Castillo-Sandoval A, Diaz-Caraballo E, Rodriguez-Guinea I, Dominguez-Lopez J. Hypoalbuminemia on admission in COVID-19 infection: An early predictor of mortality and adverse events. A retrospective observational study. Med Clin (Barc). 2021 May 7;156(9):428-436. doi: 10.1016/j.medcli.2020.12.018. Epub 2021 Jan 28. PMID 33627230
- [Result] Abumayyaleh M, Nunez Gil IJ, El-Battrawy I, Estrada V, Becerra-Munoz VM, Aparisi A, Fernandez-Rozas I, Feltes G, Arroyo-Espliguero R, Trabattoni D, Lopez-Pais J, Pepe M, Romero R, Garcia DRV, Biole C, Astrua TC, Eid CM, Alfonso E, Fernandez-Presa L, Espejo C, Buonsenso D, Raposeiras S, Fernandez C, Macaya C, Akin I; HOPE COVID-19 investigators. Does there exist an obesity paradox in COVID-19? Insights of the international HOPE-COVID-19-registry. Obes Res Clin Pract. 2021 May-Jun;15(3):275-280. doi: 10.1016/j.orcp.2021.02.008. Epub 2021 Mar 3. PMID 33741308
- [Result] Abumayyaleh M, Nunez-Gil IJ, El-Battrawy I, Estrada V, Becerra-Munoz VM, Uribarri A, Fernandez-Rozas I, Feltes G, Arroyo-Espliguero R, Trabattoni D, Lopez Pais J, Pepe M, Romero R, Ortega-Armas ME, Bianco M, Astrua TC, D'Ascenzo F, Fabregat-Andres O, Ballester A, Marin F, Buonsenso D, Sanchez-Gimenez R, Weiss C, Fernandez Perez C, Fernandez-Ortiz A, Macaya C, Akin I. Sepsis of Patients Infected by SARS-CoV-2: Real-World Experience From the International HOPE-COVID-19-Registry and Validation of HOPE Sepsis Score. Front Med (Lausanne). 2021 Oct 14;8:728102. doi: 10.3389/fmed.2021.728102. eCollection 2021. PMID 34805199
- [Result] Perez-Segura P, Paz-Cabezas M, Nunez-Gil IJ, Arroyo-Espliguero R, Maroun Eid C, Romero R, Fernandez Rozas I, Uribarri A, Becerra-Munoz VM, Garcia Aguado M, Huang J, Rondano E, Cerrato E, Rodriguez EA, Ortega-Armas ME, Raposeiras Roubin S, Pepe M, Feltes G, Gonzalez A, Cortese B, Buzon L, El-Battrawy I, Estrada V. Prognostic factors at admission on patients with cancer and COVID-19: Analysis of HOPE registry data. Med Clin (Barc). 2021 Oct 8;157(7):318-324. doi: 10.1016/j.medcli.2021.02.021. Epub 2021 May 6. PMID 34154809
- [Result] Salgado-Aranda R, Perez-Castellano N, Nunez-Gil I, Orozco AJ, Torres-Esquivel N, Flores-Soler J, Chamaisse-Akari A, Mclnerney A, Vergara-Uzcategui C, Wang L, Gonzalez-Ferrer JJ, Filgueiras-Rama D, Canadas-Godoy V, Macaya-Miguel C, Perez-Villacastin J. Influence of Baseline Physical Activity as a Modifying Factor on COVID-19 Mortality: A Single-Center, Retrospective Study. Infect Dis Ther. 2021 Jun;10(2):801-814. doi: 10.1007/s40121-021-00418-6. Epub 2021 Mar 14. PMID 33715099
- [Result] Bertaina M, Nunez-Gil IJ, Franchin L, Fernandez Rozas I, Arroyo-Espliguero R, Viana-Llamas MC, Romero R, Maroun Eid C, Uribarri A, Becerra-Munoz VM, Huang J, Alfonso E, Marmol-Mosquera F, Ugo F, Cerrato E, Fernandez-Presa L, Raposeiras Roubin S, Feltes Guzman G, Gonzalez A, Abumayyaleh M, Fernandez-Ortiz A, Macaya C, Estrada V; HOPE COVID-19 investigators. Non-invasive ventilation for SARS-CoV-2 acute respiratory failure: a subanalysis from the HOPE COVID-19 registry. Emerg Med J. 2021 May;38(5):359-365. doi: 10.1136/emermed-2020-210411. Epub 2021 Mar 16. PMID 33727235
- [Derived] Rivera-Caravaca JM, Nunez-Gil IJ, Lip GYH, Uribarri A, Viana-Llamas MC, Gonzalez A, Castro-Mejia AF, Alonso Gonzalez B, Alfonso E, Garcia Prieto JF, Cavallino C, Cortese B, Feltes G, Fernandez-Rozas I, Signes-Costa J, Huang J, Garcia Aguado M, Pepe M, Romero R, Cerrato E, Becerra-Munoz VM, Raposeiras Roubin S, Santoro F, Bagur R, Sposato L, El-Battrawy I, Lopez Masjuan A, Fernandez-Ortiz A, Estrada V, Macaya C, Marin F. Chronic Oral Anticoagulation Therapy and Prognosis of Patients Admitted to Hospital for COVID-19: Insights from the HOPE COVID-19 Registry. Int J Clin Pract. 2022 May 26;2022:7325060. doi: 10.1155/2022/7325060. eCollection 2022. PMID 35685504
- [Derived] El-Battrawy I, Longo F, Nunez Gil IJ, Abumayyaleh M, Gianesin B, Estrada V, Aparisi A, Arroyo-Espliguero R, Balocco M, Barella S, Beccaria A, Bonetti F, Casale M, De Michele E, Denotti AR, Fidone C, Fortini M, Gamberini MR, Graziadei G, Lisi R, Massa A, Marcon A, Rubinski B, Miano M, Motta I, Pinto VM, Piperno A, Mariani R, Putti MC, Quota A, Ribersani M, Marziali M, Roberti D, Rosso R, Tartaglione I, Vitucci A, Voi V, Zecca M, Romero R, Marouneld C, Fernandez-Rozas I, Espejo C, Marhaeni W, Garcia Aguado M, Cappellini MD, Perrotta S, De Franceschi L, Piga A, Forni GL, Akin I. Thalassaemia is paradoxically associated with a reduced risk of in-hospital complications and mortality in COVID-19: Data from an international registry. J Cell Mol Med. 2022 May;26(9):2520-2528. doi: 10.1111/jcmm.17026. Epub 2022 Mar 30. PMID 35355397
- [Derived] Biole C, Bianco M, Nunez-Gil IJ, Cerrato E, Spirito A, Roubin SR, Viana-Llamas MC, Gonzalez A, Castro-Mejia AF, Eid CM, Fernandez-Perez C, Uribarri A, Alfonso-Rodriguez E, Ugo F, Guerra F, Feltes G, Akin I, Fernandez-Rozas I, Blasco-Angulo N, Huang J, Aguado MG, Pepe M, Romero R, Becerra-Munoz VM, Estrada V, Macaya C. Gender Differences in the Presentation and Outcomes of Hospitalized Patients With COVID-19. J Hosp Med. 2021 Jun;16(6):349-352. doi: 10.12788/jhm.3594. PMID 34129486